CLINICAL TRIAL: NCT05354115
Title: Sample Collection for Evaluation of the Panbio™ COVID-19/ Flu A&B Rapid Panel.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDRD-H-002-P
Record Dates: First submitted 2022-04-06; First posted 2022-04-29 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Influenza A; Influenza Type B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sampling (Other): Every second participant will be instructed to blow their nose. Study personnel will then collect one nasal swab from both nostrils and two NP swabs, one from each nostril from each participant.
  Nasal samples must always be collected prior to the Nasopharyngeal sampling. A minimum of 90 Flu A positive subjects, a minimum of 90 Flu B positive subjects and a minimum of 100 SARS-CoV-2 positive subjects will be enrolled. In addition, a minimum of 385 negative subjects will be enrolled.
  Interventions: Diagnostic Test: Nasal and Nasopharyngeal Sampling of the Panbio™ COVID-19/ Flu A&B Rapid Panel

INTERVENTIONS:
Diagnostic Test: Nasal and Nasopharyngeal Sampling of the Panbio™ COVID-19/ Flu A&B Rapid Panel — Collection procedure will be a mid-turbinate nasal swab (deep nasal swab), by turning the swab five times in each nostril. After the nasal sampling, the operators will collect two nasopharyngeal swab one from each nostril of each subject.

SUMMARY:
This study is designed as a prospective, multicentric, sample collection study. The collected samples will be used for diagnostic research, product development and validation of the Panbio™ COVID-19/ Flu A&B Rapid Panel for the qualitative detection of COVID-19 antigen, Influenza A antigen (H1N1 and H3N2), and Influenza B antigen in human nasal and nasopharyngeal swabs by the study sponsor, Abbott.

DETAILED DESCRIPTION:
A minimum of 665 male and female Subjects will be prospectively enrolled at multiple clinical sites. A minimum of 90 Flu A reference positive subjects, a minimum of 90 Flu B reference positive subjects and a minimum of 100 SARS-CoV-2 reference positive subjects will be enrolled. In addition, a minimum of 385 reference-negative subjects will be enrolled. In order to meet these minimum numbers it is anticipated that approximately 2000 subjects will be enrolled in total.

Subjects should be enrolled from point of care for this study. After informed consent has been obtained, operators will collect one nasal swab from both nostrils from each Subject. Every second subject will be asked to blow their nose first and this will be recorded.

Collection procedure will be a mid-turbinate nasal swab (deep nasal swab), by turning the swab five times in each nostril.

The collected swab will be returned to a plastic tube (provided by the sponsor) and immediately (or within 15 minutes of collection) stored frozen at -80°C (or -20°C if -80°C storage is not available) for later testing with the Panbio™ Rapid Panel. Touching of the tube wall with the swab should be avoided. Nasal samples must be collected prior to the Nasopharyngeal sampling.

After the nasal sampling, the operators will collect a nasopharyngeal swab from one nostril of each subject. The NP swab will be returned to a plastic tube (provided by the sponsor) by study staff (touching the tube walls should be avoided) and immediately (or within 15 minutes of collection) stored frozen at -80°C (or -20°C if -80°C storage is not available) for later testing with the Panbio™ Rapid Panel.

A second nasopharyngeal swab, collected from the other nostril of each subject will be eluted in Universal Transport Media (UTM) and used for testing with RT-PCR protocols for Flu A, Flu B and SARS-CoV-2 as per local procedures. The remaining UTM will be labelled with Subject ID and immediately stored frozen at -80°C (or -20°C minimum). The RT-PCR methods used must have CE marking or FDA approval, with COVID-19 and Flu assay clearance for nasopharyngeal specimens and must be approved by the Sponsor. Nasopharyngeal sampling should be performed by trained healthcare professionals who routinely conduct nasopharyngeal sampling as part of their other standard of care and clinical duties.

All other aspects of the Subject's care will remain the same with no deviation from prescribed practice.

Each subject's demographic information, symptomology data, and professionally performed test result and questionnaire will be recorded on source documentation and transferred to an Electronic Data Capture system.

Samples collected in this study will be used for diagnostic research, product development and validation of the Panbio™ COVID-19/ Flu A&B Rapid Panel by the study sponsor, Abbott.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >14 years of age who are able and willing to provide written informed consent, and deemed suitable for nasopharyngeal sampling in accordance with local procedures, suspected of having a respiratory viral infection consistent with COVID-19 and/or Flu by their healthcare provider within the first five days of the onset of symptoms, and presenting at least two of the following symptoms: fever, headache, extreme tiredness, dry cough, sore throat, runny or stuffy nose, muscle aches, loss of smell, loss of taste or shortness of breath, will be prospectively enrolled.

Exclusion Criteria:

* • Subject has had a nasal or a nasopharyngeal swab taken within the last 4 hours.

  * Subject has active nose bleeds or acute facial injuries/trauma
  * Subject has received a nasal vaccine (i.e., FluMist®) within the previous five (5) days.
  * Subject is currently taking or has taken an antiviral medication-i.e., Amantadine, Rimantadine, Relenza® (Zanamivir), Tamiflu® (Oseltamivir Phosphate), and Flumadine®-for influenza within the previous thirty (30) days.
  * Subject is currently enrolled in a study to evaluate an investigational drug.
  * Subject is unwilling or unable to provide informed consent.
  * Vulnerable populations as deemed inappropriate for study by the site's PI and/or reviewing REC.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Nasal and Nasopharyngeal Sample Collection | 6 months
  The objective of this study is to collect nasal and nasopharyngeal swab specimens from individuals suspected of respiratory viral infection consistent with COVID-19 and/or Flu by their healthcare provider within the first five days of the onset of symptoms. The collected samples will be sent to the sponsor (Abbott) or central laboratory for reference testing, diagnostic research, product development and validation of the Panbio™ COVID-19/ Flu A&B Rapid Panel some of which will be used to support product registrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Urgent Care Clinical Trials Easley, Easley, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided